CLINICAL TRIAL: NCT04577794
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of GLPG3970, Administered Orally for 6 Weeks in Adult Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study Evaluating the Effects of GLPG3970 Given as an Oral Treatment for 6 Weeks in Adults With Ulcerative Colitis
Acronym: SEA TURTLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG3970-CL-210; 2020-000659-11 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Results first posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-04

CONDITIONS: Ulcerative Colitis
Keywords: Colitis; Ulcer; Moderately active ulcerative colitis; Chronic inflammatory bowel disease; Inflammatory Bowel Diseases; Digestive System Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Ulcer; Inflammatory Bowel Diseases; Digestive System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG3970 (Experimental): Participants received 400 milligrams (mg) GLPG3970 oral solution, once daily (QD) for a period of 6 weeks.
  Interventions: Drug: GLPG3970
- Placebo (Placebo Comparator): Participants received GLPG3970 matching placebo oral solution, QD for a period of 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG3970 — GLPG3970 powder and solvent for oral solution reconstituted prior to use.
  Arms: GLPG3970
Drug: Placebo — Placebo powder and solvent for oral solution reconstituted prior to use.
  Arms: Placebo

SUMMARY:
The primary objective of this study was to evaluate the effect of GLPG3970 compared to placebo on the signs and symptoms of Ulcerative Colitis (UC) in participants with moderately to severely active UC.

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented diagnosis of UC of ≥3 months. The criteria for documentation of UC diagnosis based on endoscopy will be medical record documentation, and/or a colonoscopy report dated ≥3 months before screening, which shows features consistent with UC.
2. Treatment-experienced participants with moderately to severely active disease, who have either previously demonstrated inadequate clinical response, loss of response, or intolerance to at least 1 course of standard-of-care (SoC) therapy for UC (i.e. steroids [oral or parenteral, including but not limited to prednisone, prednisolone, budesonide], 5-aminosalicylate [5- ASA] derivatives [including but not limited to mesalamine, sulfasalazine], anti-metabolites [including but not limited to azathioprine, 6 mercaptopurine, methotrexate], anti-tumor necrosis factor [TNF] agents, anti-integrins, Janus kinase [JAK] inhibitors), as confirmed by the investigator.
3. Moderately to severely active UC as determined at screening by:

   1. Centrally-read endoscopic evidence of disease activity (MCS- endoscopy subscore [ES] ≥2 OR ulcerative colitis endoscopic index of severity [UCEIS] ≥4) with a minimum disease extent of 15 cm from anal verge; AND
   2. MCS stool frequency (SF) subscore ≥1; AND
   3. MCS rectal bleeding (RB) subscore ≥1.
4. Participants currently receiving the following SoC therapies for UC are eligible providing they have been on a stable dose for the designated period of time and are anticipated to be stable throughout the study:

   1. oral corticosteroids (prednisone ≤20 mg/day or equivalent or budesonide ≤3 mg/day) stable dose for at least 2 weeks prior to first investigational product (IP) dosing.
   2. oral 5-ASA compounds (mesalamine ≤4 grams [g]/day or sulfasalazine ≤4 g/day) stable dose for at least 4 weeks prior to first IP dosing.
   3. oral thiopurines (azathioprine ≤2.5 mg/kg/day and 6-mercaptopurine 1.5 mg/kilograms [kg]/day) stable dose for at least 12 weeks prior to first IP dosing, or methotrexate ≤20 mg/week, stable dose for at least 12 weeks prior to first IP dosing.

Key Exclusion Criteria:

1. Diagnosis of Crohn's disease, indeterminate colitis, ischemic colitis, fulminant colitis, or toxic megacolon.
2. Prior surgical intervention for UC (e.g. colectomy, partial colectomy, ileostomy or colostomy) or likely requirement for surgery for UC, during the study.
3. History or evidence of incompletely resected colonic mucosal dysplasia.
4. Exhibit acute severe UC per the following criteria:

   1. bloody diarrhea ≥6/day AND
   2. any of the following signs of systemic toxicity: Body temperature (oral or tympanic) ≥37.8 degrees celsius (°C) OR Resting pulse (after 5 min seated position) >90 beats per min OR hemoglobin <105 g/L, OR erythrocyte sedimentation rate >30 millimeters per hour (mm/h); OR C-reactive protein (CRP) >30 mg/L.
5. Screening stool sample positive for ova and/or parasites, Clostridium difficile toxin, Escherichia coli, Salmonella species (spp), Shigella spp, Campylobacter spp or Yersinia spp.
6. Participant testing positive at screening for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as detected by real time polymerase chain reaction (RT-PCR), participants presenting any signs or symptoms as detected at baseline following careful physical examination (e.g. cough, fever, headaches, fatigue, dyspnea, myalgia, anosmia, dysgeusia, anorexia, sore throat, others) or reporting any signs and symptoms for the preceding 2 weeks, or participants who have been exposed to individuals with confirmed or suspected diagnosis of SARS-CoV-2 within 2 weeks prior to baseline. In addition, any other locally applicable standard diagnostic criteria may also apply to rule out SARS-CoV-2 infection.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Medical Director, Study Director — Galapagos NV
Locations (15):
- Arensia Exploratory Medicine LLC, Tbilisi, Georgia
- ARENSIA Exploratory Medicine Phase I Unit, Chisinau, Moldova
- Poland (3):
  - Centrum Medyczne PROMED, Krakow
  - Endoskopia Sp. z o.o., Sopot
  - ETG Zamosc, Zamość
- Ukraine (10):
  - I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2, Kharkiv
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - Communal Nonprofit Enterprise Kherson City Clinical Hospital n.a. Afanasii and Olga Tropini, Kherson
  - Medical Center "Harmoniya Krasy", Kyiv
  - Med Center 'Ok!Clinic+' of International Institute of Clinical Trials LLC, Kyiv
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted across 4 countries (Georgia, the Republic of Moldova, Poland, and Ukraine).
Pre-assignment Details: A total of 65 participants were screened, out of which 31 were randomized and treated.
Period: Overall Study
Arm/Group | GLPG3970 | Placebo
Started | 21 | 10
Completed | 20 | 9
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants who received at least 1 dose of investigational product (IP).
Groups:
- GLPG3970: Participants received 400 mg GLPG3970 oral solution, QD for a period of 6 weeks.
- Total: Total of all reporting groups
Arm/Group | GLPG3970 | Placebo | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (10.9) | 37.8 (5.8) | 39.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 16 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 10 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 10 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Total Mayo Clinical Score (MCS) [Mean (Standard Deviation); unit: units on a scale] — The MCS is the primary tool for assessing ulcerative colitis activity. Total MCS is the sum of 4 subscores (i.e., stool frequency, rectal bleeding, endoscopic findings, and a physician's global assessment); each rated on a scale from 0 (normal) to 3 (severe). The total MCS value ranges from 0 to 12, with higher scores indicating more severe disease.
  units on a scale | 8.5 (1.2) | 8.2 (1.3) | 8.4 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total MCS at Week 6
Description: The MCS is the primary tool for assessing ulcerative colitis activity. Total MCS is the sum of 4 subscores (i.e., stool frequency, rectal bleeding, endoscopic findings, and a physician's global assessment); each rated on a scale from 0 (normal) to 3 (severe). The total MCS value ranges from 0 to 12, with higher scores indicating more severe disease. Missing data were imputed using Rubin's multiple imputation.
Time Frame: Baseline and Week 6
Population: Full analysis set consisted of all randomized participants who received at least 1 dose of IP. Participants with available data at specified timepoint were included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 18 | 9
units on a scale | -2.6 (0.57) | -2.6 (0.85)
Statistical Analysis 1: Comparison: GLPG3970 vs Placebo; An analysis of covariance (ANCOVA) was used with a multiple imputation method to handle missing values, with treatment as fixed effect and baseline score as covariate; Test type: Superiority; p = 0.981, ANCOVA; Least square (LS) mean difference = 0.0, 90% CI 2-sided [-1.7 to 1.7], Standard Error of Mean 1.02

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-Emergent Adverse Events (TEAEs) were defined as
  * Any adverse event (AE) with an onset date on or after the IP start date and no later than 14 days after last dose of IP, or worsening of any AE on or after the IP start date.
  * Improvement or no change of any ongoing AEs on or after the IP start date are not considered treatment-emergent. If an AE was ongoing at the time of first IP intake and if there was no change or an improvement in its toxicity grade or its seriousness status, this AE was not considered as treatment-emergent.
  Serious TEAE was defined as a TEAE that
  * Resulted in death and was life-threatening;
  * Required in-patient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly / birth defect;
  * Was medically significant.
Time Frame: First dose date up to 14 days after the last dose of study drug (up to 57 days)
Population: Participants in the safety analysis set were analyzed.
Measure: Number; unit: participants
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 21 | 10
participants
  TEAEs | 11 | 3
  Serious TEAEs | 0 | 0
  TEAEs leading to death | 0 | 0
  Treatment-related TEAEs | 4 | 1
  TEAEs leading to study drug discontinuation | 1 | 0

3. Secondary Outcome: Plasma Concentration (Ctrough) of GLPG3970
Description: Ctrough was defined as plasma concentration level at the end of the dosing interval.
Time Frame: Day 15: pre-dose; Day 29: pre-dose; Day 43: pre-dose
Population: Pharmacokinetic analysis set consisted of all participants who received at least 1 dose of IP with available plasma concentration data. Participants with available plasma concentration at specified time point were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | GLPG3970
Number analyzed (Participants) | 16
nanograms per milliliter (ng/mL)
  Day 15: Pre-dose | 73.2 (145)
  Day 29: Pre-dose: number analyzed (Participants) | 15
  Day 29: Pre-dose | 55.9 (65.3)
  Day 43: Pre-dose: number analyzed (Participants) | 11
  Day 43: Pre-dose | 84.9 (107)

ADVERSE EVENTS:
Time Frame: First dose date up to 14 days after the last dose of study drug (up to 57 days)
Description: Participants in the safety analysis set were analyzed.
Arm/Group | GLPG3970 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 11/21 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG3970 (N=21) | Placebo (N=10)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 3 (4) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Blood lactate dehydrogenase decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04577794/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT04577794/SAP_001.pdf